CLINICAL TRIAL: NCT04311125
Title: Comparative Study of Minimally Invasive Surgical Approaches for Total Hip Arthroplasty: a Biochemical, Imaging and Clinical Evaluation in the Early Postoperative Period
Brief Title: Comparative Study of Minimally Invasive Surgical Approaches for Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Vasileios S. Nikolaou, Associate Professor of Orthopaedics, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Hip Osteoarthritis; Hip Arthropathy; Minimal Invasive; Anterior Approach; Tissue Injury
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- total hip arthroplasty via the mini posterior approach (Active Comparator): total hip arthroplasty via the mini posterior approach. This approach was first described by Kocher and Langenbeck and later modified by Gibson in 1950. There is a convex incision centered on the posterior rim of the major trochanter. The incision follows the curve of the buttock and at the height of the posterior lip of the major trochanter, it is peripherally oriented along the posterior outer surface of the femur. The major gluteus is divided along the muscle fibers. Guiding sutures are inserted into the tendon mass of the hip rotor muscles just prior to their origin on the major trochanter and dissected to expose and subsequently retract the posterior hip capsule.
  Interventions: Procedure: Mini posterior approach Total Hip Replacement
- THR via the anterior approach without traction table (Active Comparator): The anterior approach is a modification of the classic Smith- Peterson anterior hip approach as described by Berend et al in 2009 [7]. This approach utilizes the intermuscular plane between the tendon fascia lata and the sartorius muscle, and laterally repairs the fibers of the rectus femur to expose and enclose the anterior pubic joint. A surgical traction table may be used during surgery.
  Interventions: Procedure: Anterior approach total hip replacement without a traction table
- THR via the anterior approach with a traction table (Active Comparator): The anterior approach is a modification of the classic Smith- Peterson anterior hip approach as described by Berend et al in 2009 [7]. This approach utilizes the intermuscular plane between the tendon fascia lata and the sartorius muscle, and laterally repairs the fibers of the rectus femur to expose and enclose the anterior pubic joint. A surgical traction table may be used during surgery.
  Interventions: Procedure: Anterior approach total hip replacement with a traction table

INTERVENTIONS:
Procedure: Mini posterior approach Total Hip Replacement — Total hip replacement in patients suffering from hip osteoarthritis using the mini posterior approach
  Arms: total hip arthroplasty via the mini posterior approach
Procedure: Anterior approach total hip replacement without a traction table — Mini Anterior approach total hip replacement in patients suffering from hip osteoarthritis without the aid of a traction table
  Arms: THR via the anterior approach without traction table
Procedure: Anterior approach total hip replacement with a traction table — Mini Anterior approach total hip replacement in patients suffering from hip osteoarthritis with the aid of a traction table
  Arms: THR via the anterior approach with a traction table

SUMMARY:
Total hip arthroplasty is a method of choice for treating advanced osteoarthritis of the hip and one of the most frequent orthopedic procedures. Of all hip surgical approaches described, the tendency for minimally invasive techniques has been dominated over the last few years due to faster patient mobilization, reduced postoperative pain and need for blood transfusion. Two of the most common approaches used for minimally invasive total hip arthroplasty are: AMIS anterior approach and mini-posterior approach, which is a modification of the standard posterior approach. The purpose of this study is the biochemical, imaging and clinical evaluation of the tissue damage caused by the above-mentioned techniques of minimally invasive total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients that sign the Informed consent
* Patients aged 18 years and over who are going to undergo primary total hip arthroplasty

Exclusion Criteria:

I. Active infection II. Previous hip operation in any leg III. Any kind of operation the past 3 months IV. Obesity (BMI, Body Mass Index >30) V. Autoimmune diseases or myositis of any etiology VI. Active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Tissue damage change | Change from 6 to 24 and then 48 hours post-surgery
  Investigate and quantify at the biochemical level with all available biomarkers the extent of tissue damage caused during a hip arthroplasty between different hip surgical approaches.

SECONDARY OUTCOMES:
Imaging | Day 30 after surgery
  All patients will be subjected to imaging with a hip MRI
Clinical Tests change | Change to clinical test from Day 2 to day 15 and then day 30 post-surgery
  All patients will be monitored postoperatively for the prescribed period and data will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Orthopaedics, Athens, Attica, Greece